CLINICAL TRIAL: NCT04547504
Title: Randomized, Open-label, Controlled Phase III Trial Comparing Pembrolizumab-platinum Based Chemotherapy Combination With Pembrolizumab Monotherapy in First Line Treatment of Non-small-cell Lung Cancers (NSCLC) With PDL1 Expression ≥50%
Brief Title: PEmbRolizumab verSus chEmotherapy and pEmbrolizumab in Non-small-cell Lung Cancers (NSCLC) With PDL1 ≥ 50 %
Acronym: PERSEE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29BRC20.0159_GFPC01-2020; GFPC 01-2020 (Other: Groupe Français de Pneumo-Cancérologie)
Record Dates: First submitted 2020-08-31; First posted 2020-09-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Non-small-cell lung cancer; PDL1≥50%; advanced stage; Pembrolizumab; Chemotherapy-pembrolizumab combination
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: A national, multicenter, phase III, prospective, open label, 1:1 randomized, interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Active Comparator): Pembrolizumab
  Interventions: Drug: Pembrolizumab
- Chemotherapy-Pembrolizumab (Active Comparator): Chemotherapy and Pembrolizumab
  Interventions: Drug: Pembrolizumab and Chemotherapy drugs

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg once every 3 weeks for a maximum of 35 cycles or until disease progression, death, unacceptable toxicity, or the Investigator's or the patient's decision to stop.
  Arms: Pembrolizumab
Drug: Pembrolizumab and Chemotherapy drugs — An induction therapy followed by a maintenance therapy.
  4 induction cycles every 3 weeks associating, on the first day of each cycle:
  * Cisplatin 75mg/m² or carboplatin AUC 5mg/mL/min, pemetrexed 500mg/m² and pembrolizumab 200mg for non squamous NSCLC.
  * Carboplatin AUC 6mg/mL/min, paclitaxel 200mg/m² and pembrolizumab 200mg for squamous NSCLC.
  After the 4 induction cycles, a maintenance therapy will be possible for patients who are responding or stable:
  * Non squamous NSCLC: pembrolizumab and pemetrexed combination or either drug as monotherapy.
  * Squamous NSCLC: pembrolizumab monotherapy.
  For pembrolizumab: treatment may be continued for a maximum of 35 cycles or until disease progression, death, unacceptable toxicity, or following the Investigator's or the patient's decision to stop.
  For pemetrexed, treatment may be continued until disease progression, death, unacceptable toxicity, or following the Investigator's or the patient's decision to stop.
  Arms: Chemotherapy-Pembrolizumab

SUMMARY:
PERSEE is a French national phase 3 academic study comparing the chemotherapy-pembrolizumab combination to pembrolizumab alone as a first-line treatment for advanced NSCLC molecularly defined by a PDL1 expression ≥ 50% of tumour cells and no EGFR mutations or ALK rearrangement.

The main hypothesis is the superiority of the chemo-immunotherapy combination over mono-immunotherapy in terms of progression-free survival evaluated by an independent review committee.

One of the anticipated benefits of using the chemotherapy-pembrolizumab combination starting from the first line setting for NSCLC patients with PD L1 ≥ 50% is a reduced risk of early progression, which is known to occur with pembrolizumab monotherapy, and therefore, a better PFS.

DETAILED DESCRIPTION:
PERSEE is a french academic, prospective, randomized, controlled and open-label phase 3 study. This trial compares the combination of chemotherapy and pembrolizumab with pembrolizumab alone as first-line treatment for advanced NSCLC molecularly characterized by a PDL1 expression level ≥ 50% and no EGFR mutations or ALK rearrangement. This is a strategy trial whose primary objective is to evaluate the superiority of the chemotherapy-pembrolizumab combination over pembrolizumab using PFS as the primary endpoint as evaluated by an independent review committee.

PERSEE trial is planned to include 292 patients treated at approximately 30 GFPC-affiliated or GFPC-associated centres. After the screening period, patients will be randomized on a 1:1 basis to the Chemotherapy Immunotherapy Arm or the Immunotherapy Arm. Randomization will be stratified according to tumor histology (squamous versus non squamous) and according to the presence or absence of brain metastases. Patients enrolled in this study will receive either of the following treatment regimens:

1. Chemotherapy-Immunotherapy Arm:

   Four induction cycles once every 3 weeks associating, on the first day of each cycle:
   * Cisplatin 75 mg/m² or carboplatin area under the curve (AUC) 5 mg/mL/min, pemetrexed 500 mg/m² and pembrolizumab 200 mg for non-squamous NSCLC.
   * Carboplatin AUC 6 mg/mL/min, paclitaxel 200 mg/m² and pembrolizumab 200 mg for squamous NSCLC.

   After the 4 induction cycles, a maintenance therapy will be possible for patients who are responding or stable, as follows:
   * Non squamous NSCLC: pembrolizumab and pemetrexed combination or either drug as monotherapy (if toxicity has been identified for one of them).
   * Squamous NSCLC: pembrolizumab monotherapy.

   For pembrolizumab: treatment may be continued for a maximum of 35 cycles or until disease progression, death, unacceptable toxicity, or following the Investigator's or the patient's decision to stop.

   For pemetrexed, treatment may be continued until disease progression, death, unacceptable toxicity, or following the Investigator's or the patient's decision to stop.
2. Immunotherapy Arm:

Pembrolizumab 200 mg once every 3 weeks for a maximum of 35 cycles or until disease progression, death, unacceptable toxicity, or the Investigator's or the patient's decision to stop.

Evaluations will be performed every 6 weeks (±7 days) during the first 4 cycles in both treatment arms, then every 9 weeks (±7 days) for the first 12 months since D1 of cycle 1 and every 12 weeks (±7 days) thereafter.

Evaluations will include: tumor assessment according to RECIST v1.1, survival status, concomitant medications and AE recording. QoL/PRO questionnaires will be performed at each cycle for the first 5 cycles in both treatment arms, then every 9 weeks (±7 days) for the first 12 months since D1 of cycle 1 and every 12 weeks (±7 days) thereafter.

The length of the inclusion period is 36 months (3 years). The total study duration per patient will be a maximum of two years for the last patients included, and a maximum of five years for the first patients included (i.e. End-of-study Time Point for surviving patients)

The total study duration includes the following:

* Screening Period: up to 28 days.
* Treatment Period: up to 60 months.
* Post-study Follow up Period: until death or lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at diagnosis.
2. Histologically or cytologically confirmed NSCLC.
3. Stage IV NSCLC. Unresectable and non-eligible to radiotherapy stage III NSCLC are permitted.
4. For non-squamous NSCLCs and non-smoking squamous NSCLCs, no known activating mutations of EGFR and no ALK or ROS-1 rearrangements.
5. PD-L1 expression on ≥ 50 % of tumor cells, which will be determined locally.
6. No prior systemic treatment for lung cancer. Patients who received adjuvant therapy are eligible if the adjuvant therapy was completed at least 12 months prior to the development of metastatic disease.
7. Palliative radiotherapy completed within one day before randomization (stereotaxic or not) is authorized.
8. At least 1 target lesion in a non-irradiated area, measurable according to RECIST v1.1.
9. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1.
10. Life expectancy >12 weeks.
11. Patients with brain metastases at inclusion are accepted, provided that these metastases are asymptomatic, or symptomatic but treated (surgery or radiotherapy without or with corticosteroids ≤10 mg/day), and that they are stable on the day of inclusion.
12. No history of other malignant tumor during the previous 5 years, except for adequately treated carcinomas (in situ cervical carcinoma, basal cell carcinoma, squamous cell skin carcinoma) and low grade localized prostate cancer (Gleason <6).
13. Adequate organ function, as demonstrated by laboratory results within 7 days prior to the first administration of study treatment:

    1. Normal hepatic function: bilirubin ≤1.5 x upper limit of normal (ULN), alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) ≤2.5 x ULN or ≤5 x ULN in case of liver metastases
    2. Normal renal function: calculated creatinine clearance (CrCl, using local formula) of at least 60 mL/min for cisplatin or 45 ml/mn for carboplatin
    3. Normal hematological function: absolute neutrophil count ≥1.5 giga/L and/or platelets ≥100 giga/L, hemoglobin ≥8 g/dL
    4. Normal coagulation function: International Normalized Ratio (INR) or prothrombin time ≤1.5 x ULN and activated partial thromboplastin time (aPTT) ≤1.5 x ULN unless the patient is receiving anticoagulant therapy.
14. For patients of childbearing potential: use of an adequate method of contraception during the course of the study through 180 days after the last dose of study treatment (women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to the first administration of study treatment).

    Note: Abstinence is acceptable if this is the usual lifestyle and the patient's preferred contraception. For male subjects, male condom or abstinence are acceptable.
15. Signed informed consent to participate in the study
16. Affiliation with or benefit from French social security.

Exclusion criteria :

1. NSCLC with expression of PD-L1 <50%.
2. NSCLC with known activating mutation of EGFR or ALK or ROS-1 translocation.
3. Neuroendocrine tumor. In cases of mixed tumors, if small cell elements are present, the patient is ineligible.
4. Any previous treatment with immunotherapy regardless of the line of treatment.
5. Before the first dose of study treatment:

   1. Has received prior systemic treatment for metastatic disease (chemotherapy or targeted therapy).
   2. Had major surgery <3 weeks prior to first dose.
   3. Received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of study treatment.
6. Uncontrolled and untreated superior cava syndrome.
7. Untreated and unstable symptomatic brain metastases.
8. Leptomeningeal disease.
9. Serious concurrent conditions during the previous 6 months (severe or unstable angina pectoris, coronary or peripheral artery bypass graft of <6 months, class 3 or 4 congestive heart failure, ischemic stroke, grade ≥2 peripheral neuropathy, psychiatric or neurological disorders that may interfere with the patient's understanding of the study or with his/her informed consent.
10. Severe or non controlled systemic diseases deemed incompatible with the protocol.
11. Severe infections within 4 weeks prior to inclusion, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
12. Other previous or concomitant cancers, with the exception of basal cell carcinoma, squamous cell skin carcinoma, in situ cervical carcinoma treated, and low grade localized prostate cancer (Gleason score <6) if appropriately treated, unless the initial tumor has been diagnosed and definitively treated >5 years prior to the study, with no signs of relapse.
13. Psychological, family, social, or geographical factors that may interfere with the monitoring of the patient as defined by the protocol.
14. Any protected person (legal person protected by legal protection [guardianship, tutorship], person deprived of liberty, pregnant woman, breastfeeding woman, and minor).
15. Patients who participated in other concomitant studies unless observational and received study therapy or used an investigational device within 4 weeks prior to start of study treatment.
16. Known or suspected active autoimmune disease requiring an immunosuppressive therapy during the previous 6 months (corticosteroids or other immunosuppressive treatment). Any hormone replacement therapy (i.e. thyroxine [T4], insulin, or replacement systemic corticosteroids for adrenal or pituitary insufficiency, etc.) is not considered an immunosuppressive treatment and is authorized. Patients with hyperthyroidism or hypothyroidism who are stable under hormone replacement therapy may also be included.
17. Chronic use of immunosuppressive drugs and/or corticosteroids (>10 mg of prednisone daily). However, during the 14 days prior to randomization the use of the following is authorized:

    1. Corticosteroids as pre treatment for the administration of chemotherapy and/or for allergies or type IV hypersensitivity responses
    2. Daily prednisone (≤10 mg) as replacement therapy
    3. Inhaled or topical steroids.
18. Live-virus vaccination within 30 days of planned start of study treatment (seasonal flu vaccines that do not contain live virus are permitted).
19. Previous allogenic tissue or organ transplant.
20. History of human immunodeficiency virus (HIV) infection (positive HIV1/2 antibody test results).
21. Active hepatitis B or C.
22. Previous history of interstitial lung disease (ILD) or non infectious pneumonia (other than chronic obstructive pulmonary disease [COPD]), requiring oral or systemic steroids, current pneumonia, or anticipated ILD.
23. Known allergies or adverse reactions to the study drugs or hypersensitivity reaction to treatment with another monoclonal antibody (mAb).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) according to RECIST 1.1 assessed by blinded inependant centra review (BICR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, according to RECIST 1.1 assessed by blinded inependant centra review (BICR)

SECONDARY OUTCOMES:
Progression-free survival according to RECIST 1.1 evaluated by investigators | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Time from date of randomization until the date of first documented progression or death from any cause, whichever came first, according to RECIST v1.1 and evaluated by investigators
Progression-free survival according to iRECIST assessed by blinded inependant centra review (BICR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first assessed up to 60 months
  Time from date of randomization until the date of first documented progression or death from any cause, whichever came first, according to iRECIST assessed by blinded inependant centra review (BICR)
Objective Response Rate (ORR) | From date of first treatment administration until the date of first documented progression or death or the introduction of a new treatment, whichever came first, assessed up to 60 months
  Proportion of patients who achieved a complete response (CR) or partial response (PR) according to RECIST v1.1 from the date of first treatment administration until disease progression or the introduction of a new treatment.
Overall survival (OS) | From date of randomization until the date of death from any cause assessed up to 60 months
  Time from date of randomization until the date of death from any cause.
Duration of treatment (DOT) | From date of the first treatment administration until the date of last treatment administration, up to 60 months
  Time from the first treatment administration until the date of last treatment administration.
Duration of objective response (DOR) | From date of the first documented objective response (CR or PR) until the date of first documented progression or death from any cause, whichever came first, assessed up to 60 months
  Time from the first documented objective response (CR or PR) until the date of disease progression or death, whichever came first.
Adverse events (AE) | Up to 30 days after the last dose of study treatment for non-serious AEs. Up to 100 days or 30 days if initiating new treatment, after the last dose, for SAE.
  Proportion (%) of patients with any adverse event (AE) and number of events per treatment arm for all AEs, all serious AEs (SAEs) and all AEs of grade ≥3 according to the National Cancer Institute (NCI) Common terminology criteria for adverse events (CTCAE) v5.0 criteria.
Adverse events of special interest (AESI) | Up to 100 days or 30 days if initiating new treatment, after the last dose.
  Proportion (%) of patients with any adverse event of special interest (AESI), defined as immune-related AE (IrAE), according to the National Cancer Institute (NCI) Common terminology criteria for adverse events (CTCAE) v5.0 criteria. .
PFS in three subgroups of patients according to PD-L1 expression (50-74%, 75-100%, and 90-100%), presence or absence of brain metastasis and histology (squamous versus non squamous). | From date of randomization until the date of first documented progression or death from any cause, whichever came first, assessed up to 60 months
  Time from date of randomization until the date of first documented progression or death from any cause, whichever came first, according to RECIST v1.1
OS in three subgroups of patients according to PD-L1 expression (50-74%, 75-100%, and 90-100%), presence or absence of brain metastasis and histology (squamous versus non squamous). | From date of randomization until the date of death from any cause assessed up to 60 months
  Time from randomization until the date of death from any cause.
ORR in three subgroups of patients according to PD-L1 expression (50-74%, 75-100%, and 90-100%), presence or absence of brain metastasis and histology (squamous versus non squamous). | From date of first treatment administration until the date of first documented progression or death or the introduction of a new treatment, whichever came first, assessed up to 60 months
  Proportion of patients who achieved a complete response (CR) or partial response (PR) according to RECIST v1.1
DOR in three subgroups of patients according to PD-L1 expression (50-74%, 75-100%, and 90-100%), presence or absence of brain metastasis and histology (squamous versus non squamous). | From date of the first documented objective response (CR or PR) until the date of first documented progression or death from any cause, whichever came first, assessed up to 60 months
  Time from the first documented objective response (CR or PR) until the date of disease progression or death, whichever came first.
DOT in three subgroups of patients according to PD-L1 expression (50-74%, 75-100%, and 90-100%), presence or absence of brain metastasis and histology (squamous versus non squamous). | From date of the first treatment administration until the date of last treatment administration, assessed up to 60 months
  Time from the first treatment administration until the date of last treatment administration.
AE in three subgroups of patients according to PD-L1 expression (50-74%, 75-100%, and 90-100%), presence or absence of brain metastasis and histology (squamous versus non squamous). | Up to 30 days after the last dose of study treatment for non-serious AEs. Up to 100 days or 30 days if initiating new treatment, after the last dose, for SAE.
  Proportion (%) of patients with any adverse event (AE) and number of events per treatment arm for all AEs, all serious AEs (SAEs) and all AEs of grade ≥3 according to the National Cancer Institute (NCI) Common terminology criteria for adverse events (CTCAE) v5.0 criteria.
AESI in three subgroups of patients according to PD-L1 expression (50-74%, 75-100%, and 90-100%), presence or absence of brain metastasis and histology (squamous versus non squamous). | Up to 100 days or 30 days if initiating new treatment, after the last dose.
  Proportion (%) of patients with any adverse event (AE) and number of events per treatment arm for all AEs, all serious AEs (SAEs) and all AEs of grade ≥3 according to the National Cancer Institute (NCI) Common terminology criteria for adverse events (CTCAE) v5.0 criteria.

OTHER OUTCOMES:
Early progression rate | Up to 6 weeks from the first day of treatment
  proportion of patients with clinical and/or radiological tumor progression according to RECIST v1.1 before or at the first radiological evaluation at 6 weeks
Following of the quality of life with European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire of Cancer patients. | Up to 60 months
  The EORTC QLQ-C30 is a questionnaire with 30 questions developed to assess the quality of life of cancer patients.
  An essential aspect of the "modular" approach to QOL assessment adopted by the EORTC Quality of Life Group is the development of modules specific to tumour site, treatment modality, or a QOL dimension, to be administered in addition to the core questionnaire (EORTC QLQ-C30). Mini: 42. Maxi: 114. Hisher score mean worse outcome.
Following of the quality of life with European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire of Lung Cancer patients. | Up to 60 months
  The EORTC Study Group on Quality of Life has developed a modular system for assessing the quality of life of cancer patients in clinical trials composed of two basic elements: (1) a core quality of life questionnaire, the EORTC QLQ-C30, covering general aspects of health-related quality of life, and (2) additional disease- or treatment-specific questionnaire modules. Two international field studies were carried out to evaluate the practicality, reliability and validity of the core questionnaire, supplemented by a 13-item lung cancer-specific questionnaire module, the EORTC QLQ-LC13.The lung cancer questionnaire module comprises both multi-item and single-item measures of lung cancer associated symptoms (i.e. coughing, haemoptysis, dyspnoea and pain) and side-effects from conventional chemo- and radiotherapy (i.e. hair loss, neuropathy, sore mouth and dysphagia). Mini: 13. Maxi: 52. Higher score means worse outcome.
Following of the quality of life with European Quality of life 5 dimensions and 3 Levels | Up to 60 months
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Mini: 0. Maxi: 100. Higher score means better outcome.
Exploratory analyses to identify novel biomarkers | From date of randomization until the date of first documented progression, assessed up to 60 months
  Blood and tissue analyses to identify novel biomarkers of efficacy and resistance.
Progression-free survival 2 (PFS2) according to RECIST 1.1 | time from randomization to tumor progression on second-line therapy, or death from any cause.
  Time from randomization to tumor progression on second-line therapy, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Renaud DESCOURT, MD, Principal Investigator — Institut de Cancérologie, CHU Brest, Hôpital Morvan; Chantal DECROISETTE, MD, Principal Investigator — Medical Oncology, Centre Léon Bérard, Lyon; Christos CHOUAID, MD, PhD, Study Director — Service de pneumologie, CH intercommunal de Créteil
Locations (29):
- France (29):
  - CH du Pays d'Aix, Aix-en-Provence
  - CHU AMIENS - Hôpital Sud, Amiens
  - Chu Angers, Angers
  - CHRU de Brest, Brest
  - Centre de lutte contre le cancer - Centre François Baclesse, Caen
  - Centre Hospitalier Métropole Savoie, Chambéry
  - CH Intercommunal de Créteil, Créteil
  - CH La Roche Sur Yon - CHD Les Oudairies, La Roche-sur-Yon
  - Chu Dupuytren, Limoges
  - CH de Lorient - Hôpital du Scorff, Lorient
  - Centre Léon Berard, Lyon
  - Institut Paoli-Calmette, Marseille
  - Hôpital Européen Marseille, Marseille
  - CHU MARSEILLE_ Hopital Nord, Marseille
  - CH MEAUX, Meaux
  - APHP - Hôpital Cochin, Paris
  - CHU Bordeaux - Hôpital du Haut Levêque, Pessac
  - CH d'Annecy-genevois, Pringy
  - Centre Hospitalier de Cornouaille, Quimper
  - CHU RENNES - Hôpital Pontchailloux, Rennes
  - CHU ROUEN - Hôpital Charles Nicolle, Rouen
  - Saint Aubin Les Elbeuf, Saint-Aubin-lès-Elbeuf
  - CH La Réunion - Site Félix Guyon, Saint-Denis
  - CHU La Réunion - Groupe Hospitalier Sud, Saint-Pierre
  - SAINT-PRIEST EN JAREZ - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - Hôpital d'Instruction des Armées Toulon - Saint Anne, Toulon
  - Ch Villefranche Sur Saone, Villefranche-sur-Saône
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Descourt R, Chouaid C, Perol M, Besse B, Greillier L, Bylicki O, Ricordel C, Guisier F, Gervais R, Schott R, Auliac JB, Robinet G, Decroisette C. First-line pembrolizumab with or without platinum doublet chemotherapy in non-small-cell lung cancer patients with PD-L1 expression >/=50. Future Oncol. 2021 Aug;17(23):3007-3016. doi: 10.2217/fon-2020-1202. Epub 2021 Jun 22. PMID 34156285